CLINICAL TRIAL: NCT02115698
Title: Counteracting Age-related Loss of Skeletal Muscle Mass
Brief Title: Counteracting Age-related Loss of Skeletal Muscle Mass (CALM)
Acronym: CALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Lars Holm, PhD, MS, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-4-2013-070.3
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Sarcopenia; Muscle Loss
Keywords: Sarcopenia; Frailty; Ageing; Protein supplementation; Protein quality; Exercise training; Muscle protein turnover
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Frailty | interventions — Whey; Carbohydrates

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Heavy Resistance Training (Active Comparator): Heavy Resistance Training of the lower extremities three times weekly in combination with two daily 20 g whey protein and 10 g carbohydrate supplementations for 52 weeks.
  Interventions: Procedure: Heavy Resistance Training; Dietary Supplement: Protein Whey
- Light Intensity Training (Experimental): Home-based Light Intensity Training of the lower extremities three-five times weekly in combination with two daily 20 g whey protein and 10 g carbohydrate supplementations for 52 weeks.
  Interventions: Procedure: Light Intensity Training; Dietary Supplement: Protein Whey
- Protein Whey (Active Comparator): Two daily 20 g whey protein and 10 g carbohydrate supplementations for 52 weeks.
  Interventions: Dietary Supplement: Protein Whey
- Protein Collagen (Active Comparator): Two daily 20 g collagen protein and 10 g carbohydrate supplementations for 52 weeks.
  Interventions: Dietary Supplement: Protein Collagen
- Carbohydrate (Placebo Comparator): Two daily 30 g carbohydrate supplementations for 52 weeks.
  Interventions: Dietary Supplement: Carbohydrate

INTERVENTIONS:
Procedure: Heavy Resistance Training — Supervised Heavy Resistance Training three times weekly for 52 weeks.
  Arms: Heavy Resistance Training
Procedure: Light Intensity Training — Home-based Light Intensity Training three-five times weekly for 52 weeks.
  Arms: Light Intensity Training
Dietary Supplement: Protein Whey — Two daily 20 g whey protein and 10 g carbohydrate supplementations for 52 weeks.
  Arms: Heavy Resistance Training; Light Intensity Training; Protein Whey
Dietary Supplement: Protein Collagen — Two daily 20 g collagen protein and 10 g carbohydrate supplementations for 52 weeks.
  Arms: Protein Collagen
Dietary Supplement: Carbohydrate — Two daily 30 g carbohydrate supplementations for 52 weeks.
  Arms: Carbohydrate

SUMMARY:
Up to 66 healthy elderly individuals (at least 65 years old) are recruited as subjects. They will be recruited as a subgroup to protocol ID: H-4-2013-070.

Upon inclusion, each individual will be randomized into one of the five groups stratified according to gender (M/F) and 30s chair stand (<16 OR ≥16). The five groups are: Heavy Resistance Training (N=12), Light Intensity Training (N=12), Protein Whey (N=15), Protein Collagen (N=15) and Carbohydrate (N=12). The individuals randomized into one of the supplementation groups (Protein Whey, Protein Collagen or Carbohydrate) will be blinded to the supplement content.

Assessments will be performed at Baseline (before intervention start) and after 12 months of intervention.

The primary outcomes are measures of muscle protein synthesis rate measured as the fractional synthesis rate from Baseline to 12 months of intervention.

The hypotheses are i) that basal and protein-stimulated muscle protein synthesis rates are elevated in the exercise training groups after 12 months of intervention. ii) prolonged intake of protein of different quality will improve the muscle protein synthetic response to protein intake after 12 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, independently living
* Age at least 65 years

Exclusion Criteria:

* Subjects dependent on help/nursing etc.
* Chronic medical diseases: diabetes mellitus, clinical knee or hip osteoarthritis, other types of arthritis or connective tissue disorders, active cancer, renal diseases, severe chronic obstructive pulmonary disease, cardiac arrhythmias or known decreased left ventricular ejection fraction, lactose or gluten intolerance, chronic inflammatory bowel diseases, non-treated hyper/hypothyroidism, dementia
* Surgical diseases: Bone, muscle, tendon or joint injuries compromising participation in exercise regimens
* Implanted magnetic devices incompatible with MRi-scanning
* Weekly alcohol consumption > 21 units (1 unit equals 4 g of ethanol) for men and > 14 for women
* Medicine except acetylsalicylic acid, paracetamol, thyroid function hormones, statins in doses above 40 mg/day or if combined with subjective myalgia, ACE-inhibitors, angiotensin II blockers, beta-blockers, calciumantagonists, proton-pump inhibitors, thiazides, potassium-sparring diuretics and loop diuretics
* 1 hour of exercise weekly, except light activities such as stretching/gymnastics and bike-riding/walking as transportation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Basal overnight fasted muscle protein synthesis rate. | Baseline and 12 months
  Overnight fasting muscle protein synthesis will be measured at Baseline and after 12 months intervention by applying stable isotope amino acid tracer techniques and calculating the fractional synthesis rates.
Muscle protein synthesis rate response to protein intake from basal overnight fasted state. | Baseline and 12 months
  Change in the response of muscle protein synthesis rate to a single intake of 20 g whey protein and 10 g carbohydrate from the basal overnight fasted state from Baseline to 12 months intervention.
  Statistical analysis:
  Outcome 1 will be subtracted outcome 2 to calculate the difference FSR at baseline and 12 month respectively. The difference at baseline will be subtracted the difference at 12 month to calculate the delta difference. This delta difference will be analyzed as a modified intention-to-treat as well as per protocol, and we will test the following groups against each other using one-way analysis of variance of the relative group changes from baseline to 12 months: (1) WHEY vs. COLL vs. CARB and (2) HRTW vs. LITW vs. WHEY

SECONDARY OUTCOMES:
Muscle protein turnover molecular signaling and gene expression | Baseline and 12 months
  Muscle protein turnover regulation signaling and gene expression will be measured in the muscle tissue obtained for muscle protein synthesis measurements. Protein and protein activation status will be analysed by Western blot techniques. Gene expressions will be analysed by real time RT-PCR techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus L. Bechshoeft, MD, Principal Investigator — Bispebjerg Hospital; Lars Holm, assoc. prof., Principal Investigator — Bispebjerg Hospital; Michael Kjaer, MD, prof., Principal Investigator — Bispebjerg Hospital; Søren Reitelseder, PhD, Principal Investigator — Bispebjerg Hospital; Jacob Bülow, MD PhD stud, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Bulow J, Khakimov B, Reitelseder S, Bechshoft R, Jensen M, van Hall G, Engelsen SB, Holm L. Effect of 1-year daily protein supplementation and physical exercise on muscle protein synthesis rate and muscle metabolome in healthy older Danes: a randomized controlled trial. Eur J Nutr. 2023 Sep;62(6):2673-2685. doi: 10.1007/s00394-023-03182-0. Epub 2023 Jun 2. PMID 37266586
- [Derived] Bechshoft RL, Reitelseder S, Hojfeldt G, Castro-Mejia JL, Khakimov B, Ahmad HF, Kjaer M, Engelsen SB, Johansen SM, Rasmussen MA, Lassen AJ, Jensen T, Beyer N, Serena A, Perez-Cueto FJ, Nielsen DS, Jespersen AP, Holm L. Counteracting Age-related Loss of Skeletal Muscle Mass: a clinical and ethnological trial on the role of protein supplementation and training load (CALM Intervention Study): study protocol for a randomized controlled trial. Trials. 2016 Aug 9;17(1):397. doi: 10.1186/s13063-016-1512-0. PMID 27507236